CLINICAL TRIAL: NCT04560348
Title: Improving Mental Health by Cognitive Behavioral Intervention and Adventure Training for Chinese University Students in Hong Kong
Brief Title: Cognitive Behavioral Intervention and Adventure Training for Chinese University Students in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Jiayan Pan, Associate Professor, Hong Kong Baptist University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FRG2/14-15/090
Record Dates: First submitted 2020-09-09; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Cognitive Behavioral Therapy
Keywords: Chinese university student; mental health; adventure training
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Single group pre-posttest design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adventure-based cognitive behavioral intervention (Experimental): An adventure-based cognitive behavioral intervention program An 13-session adventure-based cognitive behavioral intervention program, including 6 lectures, 5 workshops and adventure games, and one adventure day camp (2 sessions). One session per week, 3 hours for each session. A variety of cognitive behavioral skills are taught in lectures and these skills are practiced in two groups (with appropriately 20 students in each group) in workshop to help students to apply these skills to cope with their own daily life stress. The adventure training includes a day adventure camp and five 40-minute adventure games in the beginning of each workshop. Skill briefing, case demonstration and debriefing, group sharing and discussion, in-class exercise and homework are used in the intervention program.
  Interventions: Other: adventure-based cognitive behavioral intervention

INTERVENTIONS:
Other: adventure-based cognitive behavioral intervention — The adventure-based cognitive behavioral intervention is a combination of cognitive behavioral therapy and adventure training. The intervention program is delivered in a 39-hour general education course in a public university in Hong Kong. The program includes 6 lectures, 5 workshops, 5 adventure games and an adventure day camp. Students are divided into two groups in workshop to practise CBT skills to deal with their own issues.

SUMMARY:
This study developed an adventure-based cognitive behavioral intervention program for Hong Kong university student. The program effectiveness was evaluated in reducing psychological distress and improving mental health of university students. The 3-month maintenance effect was also tested.

DETAILED DESCRIPTION:
University students are vulnerable to mental health problems due to the various challenges they have to face in university life. However, few studies have been conducted to evaluate the effectiveness of university counseling programs in Hong Kong. This project aims at developing and systematically evaluating a culturally adapted and adventure-based cognitive behavioral intervention (aCBI) program to decrease psychological distress and improve various mental health outcomes for Chinese university students in Hong Kong. The aCBI program was delivered in a form of general education course in a university setting. Single group Pre-posttest design was adopted.The program was evaluated its effectiveness in reducing psychological distress, perceived stress, depressive and anxiety symptoms, negative thoughts and negative emotions and increasing positive thoughts and positive emotions.

ELIGIBILITY:
Inclusion Criteria:

* be of Chinese nationality
* be studying in undergraduate programs at Hong Kong Baptist University (HKBU), as the aCBI program will be provided in the form of a general education course at this university
* have GHQ-12 scores of 2-10 (0-0-1-1) (i.e., mild to moderate levels of psychological distress)
* be willing to complete the entire process of the project.

Exclusion Criteria:

* have GHQ-12 scores of 0-1 (i.e., a low level of psychological distress) or 11-12 (i.e., a high level of psychological distress)
* have one or more psychosis
* have experienced severe depression with suicidal attempts/ideation in the past 3 months, as diagnosed by a psychiatrist or a clinical psychologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
General Health Questionnaire-12 | baseline: before the intervention program starts
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
General Health Questionnaire-12 | post-test: 1 month upon completion of the intervention program
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
General Health Questionnaire-12 | 3-month follow-up test: 3 months after completion of the intervention program
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress

SECONDARY OUTCOMES:
Perceived Stress Scale | baseline: before the intervention program starts
  10-item rating scale for perceived stress, scale score ranges from 0-4, with a higher score indicating a higher level of perceived stress
Perceived Stress Scale | post-test: 1 month upon completion of the intervention program
  10-item rating scale for perceived stress, scale score ranges from 0-4, with a higher score indicating a higher level of perceived stress
Perceived Stress Scale | 3-month follow-up test: 3 months after completion of the intervention program
  10-item rating scale for perceived stress, scale score ranges from 0-4, with a higher score indicating a higher level of perceived stress
Beck Depression Inventory | baseline: before the intervention program starts
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptions
Beck Depression Inventory | post-test: 1 month upon completion of the intervention program
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptions
Beck Depression Inventory | 3-month follow-up test: 3 months after completion of the intervention program
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptions
Beck Anxiety Inventory | baseline: before the intervention program starts
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Beck Anxiety Inventory | post-test: 1 month upon completion of the intervention program
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Beck Anxiety Inventory | 3-month follow-up test: 3 months after completion of the intervention program
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Automatic Thoughts Questionnaire | baseline: before the intervention program starts
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought
Automatic Thoughts Questionnaire | post-test: 1 month upon completion of the intervention program
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought
Automatic Thoughts Questionnaire | 3-month follow-up test: 3 months after completion of the intervention program
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought
Chinese Affect Scale | baseline: before the intervention program starts
  20-item rating scale for positive and negative emotions, score ranges from 1-6 for positive emotion subscale and negative emotion subscale, with a higher score indicating a higher level of positive/negative emotion
Chinese Affect Scale | post-test: 1 month upon completion of the intervention program
  20-item rating scale for positive and negative emotions, score ranges from 1-6 for positive emotion subscale and negative emotion subscale, with a higher score indicating a higher level of positive/negative emotion
Chinese Affect Scale | 3-month follow-up test: 3 months after completion of the intervention program
  20-item rating scale for positive and negative emotions, score ranges from 1-6 for positive emotion subscale and negative emotion subscale, with a higher score indicating a higher level of positive/negative emotion

CONTACTS AND LOCATIONS:
Overall Officials: Jiayan Pan, PhD, Principal Investigator — Hong Kong Baptist University

IPD SHARING:
Plan to Share IPD: No